CLINICAL TRIAL: NCT01951755
Title: An Observational Study for Safety and Efficacy of Erlotinib Beyond 1st Line in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Phase IV Study of Tarceva in Patients With Advanced Stage IIIB/ IV Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Kostas N Syrigos, Professor in Medical Oncology, University of Athens
Other Study IDs: ML27805
Record Dates: First submitted 2013-09-19; First posted 2013-09-27 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Inoperable NSCLC; TKIs
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An open-label, non randomized clinical trial of Tarceva as single agent in progressed non-small cell lung cancer patients.

DETAILED DESCRIPTION:
An observational non randomized clinical trial of Tarceva as single agent in progressed non-small cell lung cancer patients after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented diagnosis diagnosis of inoperable, locally advanced, recurrent or metastatic (Stage IIIB or IV) NSCLC.
* Patients must have evidence of disease but measurable disease is not mandatory.
* 18 years of age or older.
* ECOG Performance Status of 0-2.
* Life expectancy at least 12 weeks.
* Patients with advanced stage IIIB/ IV NSCLC who have received at least one course of standard systemic chemotherapy or radiation therapy or who are in the investigator's opinion not medically suitable for chemotherapy or radiotherapy.
* No more than 2 prior chemotherapy regimens are permissible. Patients must have recovered from any toxic effects and at least 3-4 weeks must have elapsed from the last dose and prior to registration (14 days for vinorelbine or other vinca alkaloids or gemcitabine). Patients who, in the opinion of the investigator, have fully recovered from surgery in less than 4 weeks may also be considered for the study. Patients must have recovered (CTC ≤ 1) from acute toxicities of any previous therapy.
* Granulocyte count ≥ 1.5 x 109/L and platelet count > 100 x 109/L.
* Serum bilirubin must be ≤ 1.5 upper limit of normal (ULN).
* AST and/or ALT ≤ 2 x ULN (or ≤ 5 x ULN if clearly attributable to liver metastasis.
* Serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 ml/min.
* Able to comply with study and follow-up procedures.
* For all females of childbearing potential a negative pregnancy test must be obtained within 72 hours before starting therapy.
* Patients with reproductive potential must use effective contraception.
* Written (signed) Informed Consent to participate in the study.

Exclusion Criteria:

* Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, hepatic, renal or metabolic disease).
* Prior therapy with systemic anti-tumour therapy with HER1/EGFR inhibitors (as small molecule or monoclonal antibody therapy).
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Patients are excluded if they have brain metastasis or spinal cord compression that is newly diagnosed and/ or has not yet been definitively treated with surgery and/ or radiation; previously diagnosed and treated CNS metastases or spinal cord compression with evidence of stable disease (clinically stable imaging) for at least 2 months is permitted.
* Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjogren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions. The use of contact lenses is not recommended during the study. The decision to continue to wear contact lenses should be discussed with the patient's treating Oncologist and the ophthalmologist.
* Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
* Nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced (inoperable stage IIIB or stage IV) NSCLC who had failed in platinum based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months
  Defined as the time period from the entry to the study until assessed disease progression or death

SECONDARY OUTCOMES:
Safety | Baseline, 4-6 months, 12 months, 24 months
  Adverse events and serious adverse events

OTHER OUTCOMES:
Response Rate | 4-6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: KOSTAS N SYRIGOS, MD, PhD, Study Chair — Oncology Unit University of Athens, Sotiria Hosp, 152 Mesogion Av
Locations (1):
- Oncology Unit Sotiria Hospital of Chest Diseases, Athens, Greece